CLINICAL TRIAL: NCT01119092
Title: The Effects of Talocrural Joint Mobilizations in Individuals With Diminished Dorsiflexion Range of Motion After Ankle Sprain
Brief Title: The Effects of Gentle Movements at the Ankle in Individuals With Diminished Range of Motion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Athletic Training Association Research & Education Foundation (Unknown)
Responsible Party: Jay Hertel, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14787; 14794 (Other Grant/Funding Number: National Athletic Trainers' Association Research & Education Foundation)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Lateral Ankle Sprain
Keywords: Ankle Sprain; Joint Mobilization; Manual Therapy; Range of Motion
MeSH Terms: conditions — Ankle Injuries | interventions — salicylhydroxamic acid; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham intervention plus standard treatment (Sham Comparator): This group will receive a "laying of hands" treatment in addition to standard treatment. The clinician will place his/her hands in a position to perform the AP joint mobilizations but will not actually perform them. The sham treatment will be performed 3 times and each will last a period of 60 seconds with a one minute rest in between.
  Interventions: Other: Sham ("laying of hands") intervention
- Control Group (No Intervention): This group will be individuals who suffer from the same injury but will be instructed to stretch at home 5 days a week for 2 weeks.
- Grade IV AP joint mobilization plus standard treatment (Experimental): This group will receive 3 60-second treatments of Grade IV AP joint mobilizations of the talus during each treatment session, with a one minute rest in between each treatment.
  Interventions: Other: Grade IV AP joint mobilizations

INTERVENTIONS:
Other: Sham ("laying of hands") intervention — The clinician will place his/her hands in a position to perform the AP joint mobilizations but will not actually perform them. The sham treatment will be performed 3 times and each will last a period of 60 seconds with a one minute rest in between.
  Arms: Sham intervention plus standard treatment
Other: Grade IV AP joint mobilizations — 3 60-second treatments of Grade IV AP joint mobilizations of the talus during each treatment session, with a one minute rest in between each treatment.
  Arms: Grade IV AP joint mobilization plus standard treatment

SUMMARY:
The purpose of this study is the examine the effects of gentle movements applied to the ankle joint and stretching on self-reported function, ankle motion and stiffness in individuals who have suffered from an ankle sprain within the last year and have decreased ankle motion.

DETAILED DESCRIPTION:
The purpose of this study is the examine the effects of a grade IV anterior to posterior joint mobilization and stretching on self-reported function, dorsiflexion range of motion, talar glide and stiffness in individuals who have suffered from an ankle sprain within the last year and have a 5° dorsiflexion range of motion deficit.

We will quantify range of motion with standard goniometric measures, stiffness with the use of an instrumented ankle arthrometer, talar glide with the use of the posterior talar glide test and self-reported function using the foot and ankle ability measure (FAAM) and FAAM-sport.

ELIGIBILITY:
Inclusion Criteria:

* History of a lateral ankle sprain within the last year
* Dorsiflexion range of motion deficit of 5°
* Return to full activity prior to participation in this study
* Individuals with dorsiflexion range of motion that is less than degrees of dorsiflexion.

Exclusion Criteria:

* A history of ankle surgery that involves intra-articular fixation
* Syndesmotic ankle sprain (to be ruled out based on the attending certified athletic trainers diagnosis)
* A history or signs of reflex sympathetic dystrophy
* Suffer from an acute injury in the lower extremity within the last 6 weeks
* Have received manual therapy for the ankle sprain prior to enrollment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Change in dorsiflexion range of motion | Baseline and 4 weeks
Change in posterior talar glide | Baseline and 4 weeks
Change in posterior talar translation | Baseline and 4 weeks

SECONDARY OUTCOMES:
Change in self reported function | Baseline and 4 weeks
Change in ankle stiffness | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hertel, PhD, Principal Investigator — University to Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States